CLINICAL TRIAL: NCT06811376
Title: Pilot Trial of Spiritual Care Interventions for Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Brooklyn Methodist Hospital (Other); The University of Texas Medical Branch, Galveston (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 23-10026611; R21MD017652 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor). The participant's oncologist is the care provider who is masked. This masking is needed to ensure the scientific integrity of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiritual Care Intervention #1 (Experimental): This is the experimental condition arm. Intervention details are being withheld until the trial concludes to protect the scientific integrity of the study.
  Interventions: Behavioral: Spiritual Care Intervention #1
- Spiritual Care Intervention #2 (Active Comparator): This is the active comparator condition arm. Intervention details are being withheld until the trial concludes to protect the scientific integrity of the study.
  Interventions: Other: Spiritual Care Intervention #2

INTERVENTIONS:
Behavioral: Spiritual Care Intervention #1 — Experimental
  Arms: Spiritual Care Intervention #1
Other: Spiritual Care Intervention #2 — Active Comparator
  Arms: Spiritual Care Intervention #2

SUMMARY:
This is a pilot trial of the effects of spiritual care interventions on spiritual well-being and readiness to engage in advance care planning (ACP) among black patients with advanced cancer recruited from outpatient settings to determine the feasibility of conducting a larger trial of effects of early integration of spiritual care into outpatient oncology care on patient outcomes.

DETAILED DESCRIPTION:
This will be a pilot, stratified block randomized controlled trial of the effects of healthcare chaplain services on spiritual well-being and advance care planning (ACP) among black advanced cancer patients (N=64) in outpatient settings at two medical institutions: NYP/Brooklyn Methodist Hospital (BMH) and the University of Texas Medical Branch (UTMB). The investigators will randomly assign patients in a 1:1 ratio to either the Spiritual Care Intervention #1 or Spiritual Care Intervention #2 arm of the trial. Intervention details are being withheld until the trial concludes to protect the scientific integrity of the study. Trial outcomes will be assessed at the primary endpoint, 2 months after the onset of the spiritual care intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a life-limiting, advanced cancer.
2. Identifies racially as black or African American.
3. Is fluent in English.

Exclusion Criteria:

1. Have received medical system-based spiritual care within the past 2 months.
2. Have already completed a DNR order.
3. Are too weak or cognitively impaired to engage in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Measure of Spiritual Well-Being as assessed by Functional Assessment of Chronic Illness Therapy--Spiritual Well-Being Scale [FACIT-Sp]. | 2 months
  The spiritual well-being outcome measure for this trial is the total score for the Spiritual Well-Being Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12-item Scale [FACIT-Sp-12], which has a range from 0 to 48. Higher scores mean greater spiritual well-being.
Readiness to Engage in Advance Care Planning as assessed by the Advance Care Planning Engagement Survey. | 2 months
  The readiness to engage in advance care planning outcome measure for this trial is the average score of 4 items in the 4-item version of the Advance Care Planning Engagement Survey. Each item as well as the average score of the 4 items have a range of 1 to 5. Higher scores mean greater readiness to engage in ACP.

SECONDARY OUTCOMES:
Number of individual participants who complete a DNR order. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Maciejewski, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - The University of Texas Medical Branch, Galveston, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No